CLINICAL TRIAL: NCT06267729
Title: A Phase I/II Open Label Study to Evaluate the Safety, Cellular Kinetics, and Efficacy of AZD0754, a Chimeric Antigen Receptor (CAR) T-cell Therapy Directed Against STEAP2, in Adult Participants With Metastatic Prostate Cancer: APOLLO
Brief Title: Study of AZD0754 in Participants With Metastatic Prostate Cancer
Acronym: APOLLO
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9660C00001
Record Dates: First submitted 2024-01-05; First posted 2024-02-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Prostate Cancer
Keywords: Prostate Cancer; Metastatic Prostate Cancer; mCRPC; Metastatic castration-resistant prostate cancer; CART; CAR-T; AZD0754
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Masking Description: Open-Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZD0754 (Experimental): AZD0754 monotherapy for treatment of participants with metastatic prostate cancer.
  Interventions: Biological: AZD0754
- AZD2287 (Experimental): AZD2287 is a novel imaging agent for STEAP2
  Interventions: Biological: AZD2287

INTERVENTIONS:
Biological: AZD0754 — Subjects will undergo leukapheresis to isolate peripheral blood mononuclear cells (PBMCs) to produce AZD0754. During AZD0754 production, subjects may receive bridging therapy for disease control. Upon successful generation of AZD0754 product, subjects will receive treatment with AZD0754 therapy. Study treatment will include lymphodepleting chemotherapy. After lymphodepleting chemotherapy AZD0754 is administered intravenously and patients will be required to stay at the hospital for a protocol specified monitoring period.
  Arms: AZD0754
Biological: AZD2287 — This is an Optional arm of the study, which subjects will separately consent to if they would like to participate. Subjects will receive doses of a radioactive imaging agent called AZD2287 followed by SPECT/CT imaging scans at two time points.
  Arms: AZD2287

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and antitumour activity of AZD0754 CAR T-cell therapy in participants with metastatic prostate cancer.

DETAILED DESCRIPTION:
This is a first-time in human, multi-center, open label, Phase I/II study of AZD0754 autologous CAR T-cell therapy administered intravenously to participants with metastatic prostate cancer. The study is intended to assess the safety, cellular kinetics, pharmacodynamics, preliminary efficacy, and feasibility of manufacturing AZD0754 for patients with metastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

Age

1. Participant must be 18 years or older at the time of signing the informed consent form.

   Type of Participant and Disease Characteristics
2. Participants with:

   1. A histologically confirmed diagnosis of metastatic adenocarcinoma of the prostate without known neuroendocrine differentiation or small cell features.
   2. Castration-resistant prostate cancer as defined by disease progression despite castration by orchiectomy or ongoing luteinising hormone-releasing hormone analogue. Participants receiving medical castration therapy with gonadotropin releasing hormone analogues should continue this treatment during the study.
   3. Measurable PSA >/=1 ng/mL AND
   4. Evidence of progression within 6 months prior to screening according to one of the following:

   (i) Radiographic disease progression in soft tissue based on Response Evaluation Criteria in Solid Tumours Version 1.1 criteria with or without PSA progression as per Prostate Cancer Working Group Criteria 3 (PCWG3) (ii) Radiographic disease progression in bone defined as the appearance of 2 or more new bone lesions on bone scan as per Prostate Cancer Working Group Criteria 3 (PCWG3).

   (iii) Evidence of disease progression in bone according to PSMA PET scan results in tandem with PSA progression according to PCWG3 criteria."
3. Participant has previously received a NHA (ie, abiraterone, enzalutamide, apalutamide, darolutamide) and a taxane as part of their treatment for prostate cancer (whether before or in the metastatic castration-resistant setting). Participants who are ineligible for taxanes or refuse these therapies may be enrolled at the discretion of the investigator.
4. For participants with pathogenic mutations in BRCA1 or BRCA2, they must also have received a PARP-inhibitor or be intolerant of this therapy. For participants with non-BRCA HRR deficiency disease, treatment with a PARP-inhibitor is at the discretion of the Investigator based on a risk/benefit analysis and discussion with the participant.
5. For participants who have high microsatellite instability or deficient DNA mismatch repair they must also have received at least one line of checkpoint inhibitors (ie, pembrolizumab), not be eligible for, or be intolerant to therapy as per NCCN or local treatment guidelines.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 prior to apheresis.
7. Minimum life expectancy of > 12 weeks prior to apheresis in the opinion of the Investigator
8. Adequate organ and marrow function.
9. Consent and provision of tumour material to assess STEAP2 expression and other correlative biomarkers retrospectively with pre- and post-treatment biopsies. Fresh baseline and on-treatment biopsies are required unless these are deemed medically unfeasible. If the participant is unable to undergo fresh biopsy, an archival tumour sample will be required (age of biopsy cannot be greater than 10 years).

Exclusion Criteria:

1. Participants with weight less than 39 kg
2. History of another primary malignancy except for malignancy treated with curative intent with no known active disease (≥ 2 years) before the first dose of study intervention and of low potential risk for recurrence. Such exceptions include non-melanoma cancer of the skin that has undergone curative therapy or adequately treated carcinoma in situ without evidence of disease.
3. Participants with known brain metastases.
4. Prior solid organ transplantation.
5. Active or prior documented autoimmune or inflammatory disorders. The following are exceptions to this criterion:

   1. Participants with vitiligo or autoimmune alopecia.
   2. Participants with autoimmune hypothyroidism (eg, following Hashimoto thyroiditis) stable on hormone replacement.
   3. Any chronic inflammatory or autoimmune skin condition that does not require systemic therapy.
   4. Participants without active disease in the last 5 years may be included, but only after consultation with the Sponsor.
   5. Participants with coeliac disease controlled by diet alone.
6. Stroke, intracranial haemorrhage, or seizure within 6 months of apheresis.
7. Cardiac arrhythmias, (such as multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia), which are symptomatic or require treatment (Common Terminology Criteria for Adverse Events [CTCAE] Grade 3) unless controlled by pacemaker (discussion with the Study Physician required); symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia.
8. Investigator judgement of one or more of the following:

   1. Mean resting corrected QT interval > 470 ms, obtained from triplicate electrocardiograms (ECGs) performed at screening.
   2. History of QT prolongation associated with other medications that required discontinuation of that medication, or any current concomitant medication known to prolong the QT interval and be associated with Torsades de Pointe.
   3. Congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first-degree relatives.
9. Uncontrolled intercurrent illness including, but not limited to, ongoing or active known infection, cardiomyopathy of any aetiology, symptomatic congestive heart failure defined by New York Heart Association class ≥ 3), interstitial lung disease, uncontrolled hypertension, uncontrolled diabetes mellitus, unstable angina pectoris, history of myocardial infarction within the past 6 months prior to apheresis, known bleeding diathesis such as haemophilia, von Willebrand disease, etc.
10. Active, uncontrolled epilepsy. Participants without active/uncontrolled epilepsy in the last 5 years may be included.
11. Persistent toxicities (CTCAE Grade ≥ 2) caused by previous anticancer therapy, excluding alopecia. Participants with irreversible toxicity that is not reasonably expected to be exacerbated by study intervention may be included (eg, hearing loss) after consultation with the Study Physician or Medical Monitor. Participants with Grade 2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician or Medical Monitor.
12. Seropositive for human immunodeficiency virus (HIV).
13. Active hepatitis C infection (HCV). Participants testing positive for HCV antibody are eligible only if the polymerase chain reaction is negative for HCV RNA.
14. Participants with hepatitis B virus (HBV) may be included under the following circumstances:

    1. Negative for hepatitis B surface antigen (HbsAg) and positive for anti-HBc antibody
    2. Positive for HbsAg, but for > 6 months have had normal transaminases and HBV DNA levels between 0 - 2000 IU/mL (inactive carrier state) and willing to start and maintain antiviral treatment for at least the duration of the study.
    3. HBV DNA levels > 2000 IU/mL but on prophylactic antiviral treatment for the past 3 months and will maintain the antiviral treatment during the study.
15. Local requirements for the testing for infectious diseases and exclusions of applicable participants should be followed per local regulations.

    Prior/Concomitant Therapy
16. Participants may not receive full-dose long-acting oral (eg, warfarin) or parenteral anticoagulants or thrombolytic agents for therapeutic (as opposed to prophylactic) purpose from the time of informed consent to 28-days post infusion of AZD0754. Use of short acting direct oral anticoagulants (eg, rivaroxaban) for therapeutic and prophylactic purposes are permitted.
17. Received the following:

    1. Major surgery within 2 weeks prior to apheresis, or planned major surgery within 4 weeks of the study treatment administration (Note: participants with planned surgical procedures to be conducted under local anaesthesia may participate after discussion with the Sponsor).
    2. Corticosteroids (except inhaled corticosteroids) or other immunomodulators (including interleukins, interferons, and thymosins) of systemic therapeutic dose, and systemic corticosteroids at doses exceeding 10 mg/day of prednisone or equivalent < 7 days prior to apheresis.
18. Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy targeted therapy, biologic therapy, tumour embolisation, or monoclonal antibodies, investigational product) within 5 half-lives or ≤ 21 days (whichever is shorter) prior to apheresis. Radiotherapy within 14 days. However, if the radiation portal covered ≤ 5% of the bone marrow reserve, the participant is eligible irrespective of the end date of radiotherapy. If sufficient washout time has not occurred due to the schedule or PK properties of an agent, a longer washout period will be required, as agreed by AstraZeneca and the Investigator.
19. Any concurrent anticancer treatment with the following exceptions:

    1. Protocol-defined LDC
    2. Hormonal therapy for non cancer-related conditions (eg, hormone replacement therapy)
    3. Androgen deprivation therapy with a luteinising-hormone replacement hormone agonist/antagonist is required if needed to maintain testosterone level in the castration range (levels < 50 ng/dL) and should be continued (unless bilateral orchiectomy) throughout the trial. Following apheresis, bridging therapy is permitted (if required) as outlined in Section 6.1.2
20. Participants should not have received any live vaccines within 30 days prior to apheresis. Participants can receive coronavirus (COVID)-19 vaccines, at the discretion of the Investigator, following a benefit/risk evaluation for the individual participant and in accordance with local rules and regulations and vaccination guidelines. Note: If a COVID-19 vaccine is administered, it should ideally be done at least one week prior to LDC or after completion of the DLT period.

    Prior/Concurrent Clinical Study Experience
21. Prior treatment with a CAR-T therapy directed at any target or any therapy that is targeted to STEAP2.
22. Participants with a known life-threatening allergy, hypersensitivity, or intolerance to AZD0754 or any of the excipients of the product, including dimethylsulfoxide.

In addition to the above, the following exclusion criteria is applicable for study participants in Australia:

- Participants with human T-lymphotropic virus (HTLV).

Ages: 18 Years to 130 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male Participants
Enrollment: 60 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2026-11-24 (Estimated); Study Completion 2026-11-24 (Estimated)

PRIMARY OUTCOMES:
Incidence of participants with Dose-limiting Toxicity (DLTs)/DLT-like events, Adverse Events (AEs), including Adverse Events of Special Interest (AESIs) and Serious Adverse Events (SAEs). | Through study completion, an average of 2 years
  Determine if treatment with AZD0754 is safe and tolerable through assessment of DLTs/DLT-like events, AEs, AESIs, SAEs, and changes from baseline in laboratory parameters, vital signs, and ECGs.

SECONDARY OUTCOMES:
Prostate-specific antigen (PSA) response rate - PSA50 | Through study completion, an average of 2 years
  PSA50 response rate is defined as the proportion of participants achieving a ≥ 50% decrease in PSA from baseline to the lowest post-baseline PSA result, confirmed by a second consecutive PSA assessment at least 3 weeks later.
PSA response rate - PSA90 | Through study completion, an average of 2 years
  PSA90 response rate is defined as the proportion of participants achieving a ≥ 90% decrease in PSA from baseline to the lowest post-baseline PSA result, confirmed by a second consecutive PSA assessment at least 3 weeks later.
Duration of PSA Response (DoPSA50, DoPSA90) | Through study completion, an average of 2 years
  Time from the date of first documented PSA50 and PSA90 until the date of documented PSA progression or death due to any cause in the absence of PSA progression.
Durable PSA Response Rate (DRRPSA50, DRRPSA90) | Through study completion, an average of 2 years
  Percentage of participants who have a confirmed PSA50 and PSA90 response with a duration of at least 6 months.
Time to PSA Response (TTPSA50, TTPSA90) | Through study completion, an average of 2 years
  Time from AZD0754 infusion date until the date of the first documented PSA50 and PSA90 response.
Time to PSA Progression (TTPSAP50, TTPSAP90) | Through study completion, an average of 2 years
  Time from the date of first documented PSA50 and PSA90 response until the date of documented PSA progression.
Best Overall Response (BOR) | Through study completion, an average of 2 years
  Best overall radiological visit response the participant achieves per RECIST V1.1 and PCWG3.
Objective Response Rate (ORR) | Through study completion, an average of 2 years
  Percentage of participants with a confirmed Complete Response (CR) or Partial Response (PR).
Time to Response (TTR) | Through study completion, an average of 2 years
  Time from AZD0754 infusion date until date of first documented evidence of CR or PR.
Duration of Response (DoR) | Through study completion, an average of 2 years
  Time from the date of first documented evidence of CR or PR until date of first documented disease progression or death.
Durable Response Rate (DRR) | Through study completion, an average of 2 years
  Percentage of participants who have a confirmed response (CR/PR) with a duration of at least 6 months.
Disease Control Rate (DCR) | 12 and 24 weeks after AZD0754 infusion
  Percentage of participants who have a confirmed CR, PR, or Stable Disease (SD) for at least 11 and 23 weeks after AZD0754 infusion.
Percentage change in tumor size | Through study completion, an average of 2 years
  Percentage change in tumor size from baseline per RECIST V1.1 and PCWG3.
Radiographic Progression-free Survival (rPFS) | Through study completion, an average of 2 years
  Time from AZD0754 infusion until date of objective disease progression according to RECIST V1.1 and PCWG3 criteria.
Overall Survival (OS) | Through study completion, an average of 2 years
  Time from AZD0754 infusion until death due to any cause
Time from AZD0754 Infusion to the first Symptomatic Skeletal-related Events (SSRE) | Through study completion, an average of 2 years
  Time from AZD0754 Infusion to the first Symptomatic Skeletal-related Event (SSRE).
Pharmacokinetics - maximum observed serum concentration (Cmax) of AZD0754 | Through study completion, an average of 2 years
  Maximum observed serum concentration
Pharmacokinetics - time taken to reach maximum serum concentration (Tmax) of AZD0754 | Through study completion, an average of 2 years
  Time taken to reach maximum serum concentration
Pharmacokinetics - Last measurable serum concentration (Clast) of AZD0754 | Through study completion, an average of 2 years
  Last measurable serum concentration
Pharmacokinetics - time of last measurable serum concentration (Tlast) of AZD0754 | Through study completion, an average of 2 years
  Time of last measurable serum concentration
Pharmacokinetics - Exposure of AZD0754 | Through study completion, an average of 2 years
  Area Under the concentration time curve
Biomarker - STEAP2 expression in Tumor | Through study completion, an average of 2 years
  Investigate STEAP2 expression in tumor as measured by IHC.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (11):
  - Research Site, Duarte, California
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Westwood, Kansas
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Hackensack, New Jersey
  - Research Site, New York, New York
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
- Research Site, East Melbourne, Australia
- Research Site, Pamplona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/